CLINICAL TRIAL: NCT05709275
Title: Hypoplastic Left Heart Syndrome: Subendocardial Viability After Norwood Palliation
Acronym: HLHS
Status: Terminated | Type: Observational
Why Stopped: early suspension of the study
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Antonio Saracino, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: HLHS
Record Dates: First submitted 2023-01-10; First posted 2023-02-02 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Hypoplastic Left Heart Syndrome
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This project has several objectives ranging from clinical data analysis to computational simulations as listed below:

1. Retrospective review of all patients with HLHS treated surgically and followed medically at the IRCCS Policlinico San Donato aiming to assess the SEVR after each step of Norwood palliation to analyze its influences on:

   * Mortality;
   * Occurrence of adverse events;
   * Outcome of the three-staged palliation;
2. Creation of a prospective registry that will enroll all patients surgically treated for HLHS at the IRCCS Policlinico San Donato.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (age ≤18 years) with the diagnosis of hypoplastic left heart syndrome who underwent the Norwood palliation at the IRCCS Policlinico San Donato.

Exclusion Criteria:

* Patients with any type of atrioventricular discordance.
* Pediatric patients (age ≤18 years) with the diagnosis of hypoplastic left heart syndrome who underwent the Norwood palliation at the IRCCS Policlinico San Donato before March 2019.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with HLHS treated surgically and followed medically at the IRCCS Policlinico San Donato
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Mortality during the hospital stay and after the discharge | 5 year
  death, cardiovascular arrest

SECONDARY OUTCOMES:
Number of adverse events registered during the follow-up. | 5 year
  Patients will be followed prospectively with their normal routine cardiological follow-up for 5 years

OTHER OUTCOMES:
Number of adverse events at the three-staged palliation (short and long-term mortality) | 5 year
  Patients will be followed prospectively with their normal routine cardiological follow-up aiming to capture adverse events and clinical status.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato, Milano, Italy

IPD SHARING:
Plan to Share IPD: No